CLINICAL TRIAL: NCT03258411
Title: Comparison of The Short Term Effects of Different Palatal Expanders Using CBCT.
Brief Title: Evaluation Of Different Rapid Orthodontic Expansion Devices
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Najla Alhamdani, Master degree student, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBRPE
Record Dates: First submitted 2017-07-22; First posted 2017-08-23 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Cross Bite
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Haas group (H) (Active Comparator): Rapid Expansion of palatal suture device: tooth-tissue supported expander (Haas (H)).
  Interventions: Device: Rapid Expansion of palatal suture
- Hyrax (Hx) (Active Comparator): Rapid Expansion of palatal suture device: tooth anchored expander (Hyrax (Hx)).
  Interventions: Device: Rapid Expansion of palatal suture
- Miniscrew-supported (MHx) (Active Comparator): Rapid Expansion of palatal suture device: bone anchored expander (Temporary anchorage devices(miniscrew)-supported (MHx))
  Interventions: Device: Rapid Expansion of palatal suture

INTERVENTIONS:
Device: Rapid Expansion of palatal suture

SUMMARY:
Evaluating and comparing the short term effects of different palatal expanders on the amount of palatal expansion and buccal tipping of posterior teeth.

Hypothesis:

H0: There is no difference in the short term effects between the different palatal expanders.

H1: There is a significant difference in the short term effects between the different palatal expanders.

ELIGIBILITY:
Inclusion Criteria:

* Non-syndromic adolescent patients.
* Patients in need for palatal expansion treatment.
* Average face height.
* No previous orthodontic treatment.

Exclusion Criteria:

* Syndromic adolescent patients.
* Patients not in need for palatal expansion treatment.
* Non-average face height.
* Previous orthodontic treatment.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2015-02-10 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Amount of skeletal and dental expansion | 3 months
  These are linear measurements which will be measured in millimetres in the first and the second cone beam computed tomography images and the difference will be calculated.
Amount of dental inclination | 3 months
  These are angular measurements which will be measured in degrees in the first and the second cone beam computed tomography images and the difference will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Faculty of Dentistry, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mosleh MI, Kaddah MA, Abd ElSayed FA, ElSayed HS. Comparison of transverse changes during maxillary expansion with 4-point bone-borne and tooth-borne maxillary expanders. Am J Orthod Dentofacial Orthop. 2015 Oct;148(4):599-607. doi: 10.1016/j.ajodo.2015.04.040. PMID 26432315
- [Background] Lagravere MO, Carey J, Heo G, Toogood RW, Major PW. Transverse, vertical, and anteroposterior changes from bone-anchored maxillary expansion vs traditional rapid maxillary expansion: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2010 Mar;137(3):304.e1-12; discussion 304-5. doi: 10.1016/j.ajodo.2009.09.016. PMID 20197161